CLINICAL TRIAL: NCT00972647
Title: Radiation Exposure Using Laser Guided Fluoroscopy in Various Orthopaedic Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of personnel
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Montri D. Wongworawat, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 59130
Record Dates: First submitted 2009-08-20; First posted 2009-09-07 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Fractures
Keywords: fracture; fixation; fluoroscopy; laser; radiation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unguided (No Intervention): Fluoroscopy images taken without laser beam guidance
- Laser guided (Experimental): Fluoroscopy images taken with laser beam guidance
  Interventions: Procedure: Laser beam guidance

INTERVENTIONS:
Procedure: Laser beam guidance — Using the laser centralizing beam to assist in position the body part prior to fluoroscopic imaging
  Arms: Laser guided

SUMMARY:
Introduction: The orthopaedic surgeon is frequently exposed to ionizing radiation, especially during intraoperative fluoroscopy. It is expected that using a laser guided fluoroscopy technique, which should improve accuracy of radiography, should also reduce the amount of time of exposure to radiation. Finally, the literature appears controversial in this matter with no clear conclusions that could be drawn from such.

Hypothesis: The test hypothesis is that the use of the laser-aiming device for fluoroscopy in several orthopaedic procedures will reduce the exposure of the patient and the surgeon to the damaging effects of radiation. The null hypothesis then states that there will be no difference in exposure to radiation between the group using the laser device and the group not using the apparatus.

Methods: A prospective randomized controlled trial will be performed in which patients undergoing fluoroscopy will be randomly allocated to two groups. One group will undergo imaging with use of the device throughout the procedure and the other group will undergo radiation without the laser guided device. Number and time of exposure will be recorded for each procedure. It is of the utmost importance that the complexity of the procedures remains relatively similar. It is believed that a good measure of complexity is the surgical time. Therefore, any procedures that are statistically similar from a set mean (p > 0.05) would be included into the study. It is also important that one or two surgeons with similar expertise and years of experience perform the surgeries to avoid confounding factors. It is expected that throughout the duration of the study (8 weeks) 50-100 cases would be reported which would produce statistically significant results. The results will be analyzed by calculating confidence intervals and differences between means of continuous data and significance levels by the Student's t test. Statistical significance will be set to P < 0.05.

Risks and Benefits: This study involves minimal risk. The use of the laser guide will not increase or introduce any risks other than the associated inherent surgical risks. The risks usually associated with this type of studies concern breach of confidentiality. To reduce this risk, research numbers will be assigned to subjects' data collected during the procedure, whose personal information will be found in another password-protected database.

This study will help the investigators to investigate a technique that may help reduce the amount of time that a patient is exposed to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractures requiring surgery with fluoroscopic assistance

Exclusion Criteria:

* Patients with fractures treated without surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Duration of radiation exposure | 1 to 12 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Montri D Wongworawat, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States